CLINICAL TRIAL: NCT00694005
Title: Phase IV Study of the Choice of Optimal Strategy for Bifurcation Lesions With Normal Side Branch
Brief Title: Choice Of Optimal Strategy For Bifurcation Lesions With Normal Side Branch
Acronym: CROSS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-0185
Record Dates: First submitted 2008-06-05; First posted 2008-06-09 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease
Keywords: stent; bifurcation; balloon angioplasty
MeSH Terms: conditions — Coronary Artery Disease | interventions — Sirolimus; Paclitaxel; zotarolimus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bifurcation stent techniqe (Active Comparator): cross over stenting without kissing balloon angioplasty "leave alone"
  Interventions: Procedure: without kissing balloon angioplasty "leave alone"
- bifurcation stent technique (Experimental): kissing balloon angioplasty
  Interventions: Procedure: kissing balloon

INTERVENTIONS:
Procedure: kissing balloon — simultaneous kissing balloon angioplasty during drug-eluting stent implantation for bifurcation coronary lesions
  Other Names: Sirolimus, Paclitaxel, Zotarolimus and Everolimus stents
  Arms: bifurcation stent technique
Procedure: without kissing balloon angioplasty "leave alone" — simultaneous kissing balloon angioplasty during drug-eluting stent implantation for bifurcation coronary lesions
  Other Names: sirolimus, zotarolimus, paclitaxel, and everolimus stents
  Arms: bifurcation stent techniqe

SUMMARY:
Few data are available about the late patency of side branches in association with the currently used stent types and implantation techniques.

DETAILED DESCRIPTION:
Among the bifurcation type, bifurcation lesion without significant side branch stenosis (<50%) usually did not require side branch stenting, but owing to several putative mechanism including dissection, thrombosis formation, embolization of plaque debris, ostial compromise by displaced stent strut, and snow plow effect, the side branch might be compromised. In this situation, the strategy to achieve optimal results has not been reported. Recently, FFR study showed that most jailed side branch (vessel size >2.0 mm. DS>50%) after main branch stenting did not have functional significance. We compared strategies with or without routine kissing balloon dilatation for less than 50% stenosis after simple DES crossing for bifurcation lesions (bifurcation type 1.1.0, 1.0.0, and 0.1.0 according to Medina classification) with serial change of FFR measurement.

ELIGIBILITY:
Inclusion Criteria:

* Clinical

  * Patients with angina and documented ischemia or patients with documented silent ischemia
  * Patients who are eligible for intracoronary stenting
  * Age >18 years, <75 ages
* Angiographic

  * De novo lesion located in a major bifurcation point with the MEDINA classification type 1.1.0, 1.0.0, or 0.1.0
  * Main vessel : >= 2.5 mm in vessel size, >= 50% in diameter stenosis and =< 50 mm in lesion length by visual estimation, in which the lesion is covered with =< 2 stents
  * Side branch :>= 2.0 mm in vessel size and < 50% diameter stenosis by visual estimation

Exclusion Criteria:

* History of bleeding diathesis or coagulopathy
* Pregnant
* Known hypersensitivity or contra-indication to contrast agent, heparin, sirolimus, paclitaxel and zotarolimus
* Limited life-expectancy (less than 1 year) due to combined serious disease
* ST-elevation acute myocardial infarction =< 2 weeks
* Characteristics of lesion:

  * Left main disease
  * In-stent restenosis
  * Graft vessels
  * TIMI flow =< grade 2 in the side branch
  * Chronic total occlusion
* Renal dysfunction, creatinine >= 2.0mg/dL
* Contraindication to aspirin, clopidogrel or cilostazol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2008-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Diameter stenosis at 8-month follow-up between the kissing balloon inflation and leave alone strategy | 8 months
  8 month after PCI

SECONDARY OUTCOMES:
Incidence of side branch jail after main vessel stenting according to the stent type used | Day 1
  Day 1 (24 hours after the index procedure)
Angiographic reocclusion rate of side branch | 8 months
  8month after PCI
Angiographic restenosis rate of side branch and the main vessel | 8 months
  8month after PCI
Late loss of side branch and the main vessel between angiography- and FFR-guided side branch procedure | 8 months
  8month after PCI
Angiographic reocclusion, restenosis rate and late loss of the side branch according to the DES type | 8 months
  8month after PCI
Angiographic reocclusion, restenosis rate and late loss of the side branch according to bifurcation angle and bifurcation type | 8 months
  8month after PCI
Composite of major cardiac adverse events (MACE) including death, MI, stent thrombosis and target vessel revascularization | 2 years
FFR of the side branch at post-procedure and at follow-up | Day 1, 8 months
  Day 1 (immediately after the index procedure)and 8month after PCI
Incidence of peri-procedural cardiac enzyme elevation | Day 1
  Day 1 (24 hours after the index procedure)
Fluoroscopic time | Day 1
  Day 1 (immediately after the index procedure)
Procedure time | Day 1
  Day 1 (immediately after the index procedure)
Amount of contrast agent | Day 1
  Day 1 (immediately after the index procedure)
Number of used stents | Day 1
  Day 1 (immediately after the index procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (11):
- South Korea (11):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Busan Saint Mary's Hospital, Busan
  - Cheongju Saint Mary's Hospital, Cheongju-si
  - Chungnam National University Hospital, Daejeon
  - Kyungsang University Hospital, Jinju
  - Hallym University Sacred Heart Hospital, Pyeongchon
  - Catholic University, Kangnam St. Mary's Hospital, Seoul
  - Hallym University Sacred Heart Hospital, Seoul
  - Aju University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Kangwon University Hospital, Wŏnju